CLINICAL TRIAL: NCT05213364
Title: Dengue Vaccine Hesitancy and Acceptance in Endemic Regions of Argentina: Impact of Communication Strategies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundacion GESICA (Other)
Responsible Party: Sponsor
Other Study IDs: Dengue_VaxHes
Record Dates: First submitted 2022-01-26; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Dengue
Keywords: Vaccine Hesitancy
MeSH Terms: conditions — Dengue; Vaccination Hesitancy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Among all arboviruses, Dengue (DEN) is the vector borne disease with the highest burden worldwide. Around 390 million infections per year are estimated, of which around 96 million are clinically apparent.

Since its re-emergence in 1998 in Argentina, DEN has shown an epidemic behavior affecting mainly the northern and central regions in which the circulation of serotypes has been heterogeneous. The last significant outbreak was registered between the end of 2019 and the beginning of 2020..

Vaccine development for DEN prevention has been a long and challenging journey. The only vaccine that has reached registration to date is a recombinant attenuated tetravalent vaccine (Dengvaxia, Sanofi Pasteur) showing an efficacy against virological confirmed DEN infection of 36.6% (4.2-61.4) in seronegative subjects at baseline and 77.9% (65.1-86.0) in seropositive. However, this vaccine has not been pre qualified by the World Health Organization. New dengue vaccines are in advanced stages of development worldwide. At least three vaccines are in advanced stages of development including one produced by Takeda, the Butantan Institute and the Merck, Sharp & Dohme development.

The implementation of a vaccination strategy in Argentina could be a health-relevant approach. However, the best way to implement this requires prior information describing and investigating numerous aspects of vaccination including acceptability.

A systematic review of two acceptability surveys showed an acceptability of 77% to 86% but in countries with endemic DEN at time of the surveys.

It is possible that in Argentina, the introduction to the regular calendar, for use in specific regions with a high and periodic burden of disease, of highly effective and safe DEN vaccines will be considered. However, to our knowledge, we do not have available evidence of the potential acceptability of these vaccines.

The main objectives of this research will be:

To evaluate the acceptability of a DEN vaccine in potential target populations in regions of high burden of disease in Argentina.

Describe main determinants of and barriers to DEN vaccine acceptability in regions of high burden of disease in Argentina.

Identify information and intervention needs to design and implement communication strategies that have a positive impact on the acceptability of a DEN vaccine.

ELIGIBILITY:
Inclusion Criteria:

* People who express willingness to participate and who are residents of communes with a high burden of Dengue disease.

Exclusion Criteria:

* Persons who do not give informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18 years or older, residing in one of the three districts with the highest burden of NDD in Argentina who provide written informed consent to participate in the survey.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who express acceptability to the DEN vaccine. | Baseline (time 0)
Proportion of subjects who express acceptability to the DEN vaccine. | At 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Angeleri, MD, Study Chair — Fundación GESICA

IPD SHARING:
Plan to Share IPD: No